CLINICAL TRIAL: NCT00080327
Title: A Placebo-Controlled Study of Three Doses of Aripiprazole in Patients With Acute Schizophrenia
Brief Title: Study of Three Doses of Aripiprazole in Patients With Acute Schizophrenia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Development & Commercialization, Inc. (Industry)
Collaborators: Otsuka America Pharmaceutical (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CN138-113 ST
Record Dates: First submitted 2004-03-26; First posted 2004-03-30 (Estimated); Last update posted 2013-11-11 (Estimated); Status verified 2008-08

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — Aripiprazole

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (4):
- 1 (Active Comparator)
  Interventions: Drug: Aripiprazole
- 2 (Active Comparator)
  Interventions: Drug: Aripiprazole
- 3 (Active Comparator)
  Interventions: Drug: Aripiprazole
- 4 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Aripiprazole — Tablets, Oral, 2mg, Once daily, 6 weeks.
  Other Names: Abilify
  Arms: 1
Drug: Aripiprazole — Tablets, Oral, 5mg, Once daily, 6 weeks.
  Other Names: Abilify
  Arms: 2
Drug: Aripiprazole — Tablets, Oral, 10mg, Once daily, 6 weeks.
  Other Names: Abilify
  Arms: 3
Drug: Placebo — Tablets, Oral, 0mg, Once daily, 6 weeks.
  Arms: 4

SUMMARY:
A study to evaluate three doses of aripiprazole versus placebo in patients with an acute episode of schizophrenia

ELIGIBILITY:
Inclusion Criteria:

* Men and women, ages 18 and older, with a worsening of schizophrenia symptoms over the past three months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 370
Dates: Start 2003-11; Primary Completion 2004-09 (Actual); Study Completion 2004-09 (Actual)

PRIMARY OUTCOMES:
Change at endpoint in schizophrenia rating scale

SECONDARY OUTCOMES:
Clinical Global Improvement scale at endpoint and time to response

CONTACTS AND LOCATIONS:
Locations (1):
- Bristol-Meyers Squibb Call Center, Wallingford, Connecticut, United States